CLINICAL TRIAL: NCT02977156
Title: A Phase I Dose Escalation Trial Evaluating the Impact of an in Situ Immunization Strategy With Intra-Tumoral Injections of Pexa-Vec in Combination With Ipilimumab in Metastatic / Advanced Solid Tumors With Injectable Lesions.
Brief Title: Immunization Strategy With Intra-tumoral Injections of Pexa-Vec With Ipilimumab in Metastatic / Advanced Solid Tumors.
Acronym: ISI-JX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET14-035 (ISI-JX)
Record Dates: First submitted 2016-11-25; First posted 2016-11-30 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Tumor; Advanced Tumor
Keywords: Injectable lesion; Intra-tumoral injection
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination PexaVec + Ipilimumab (Experimental): * PEXA-VEC (Pexastimogene devacirepvec): Oncolytic live replicating virus, Recombinant vaccinia virus GM-GCF of Classe 1, administered by Intra-tumoral injection with fixed-dosage regimen of 1x109 pfu (9.0 Log pfu)/ injection. Up to 5 IT injections, at Week 1 Day 1, Week 3 Day 1, Week 5 Day 1 and Week 9 Day 1, and one additional IT treatment allowed in case of disease progression following a documented objective response at W12. Provided by Transgene.
  * IPILIMUMAB: Anti-CTLA-4 monoclonal antibody (IgG1k) produced in CHO cells by recombinant DNA technology, administered by Intra-tumoral injection. Up to 4 IT injections at Week 3 Day 1, Week 5 Day 1 and Week 9 Day 1, and one additional IT treatment allowed In case of disease progression following a documented objective response at W12. Four dose levels of ipilimumab will be tested in dose escalation step: 2.5mg, 5mg, 7.5mg, 10mg, 20mg or 40 mg.
  Interventions: Biological: Pexa-Vec; Drug: Ipilimumab

INTERVENTIONS:
Biological: Pexa-Vec — IT Injections will be performed by a radiologist using imaging-guidance, ultrasound or computed tomography (CT). The dose to be injected could be divided between 1 to 5 tumor lesions.
  Other Names: JX-594; TG6006; VAC GM-CSF
Drug: Ipilimumab — IT Injections will be performed by a radiologist using imaging-guidance, ultrasound or computed tomography (CT). The dose to be injected could be divided between 1 to 5 tumor lesions.
  Other Names: Yervoy®

SUMMARY:
The success of anti-CTLA4 therapy has inaugurated a paradigm shift in oncology where drugs target the immune system rather than cancer cells in order to stimulate the anti-tumor immune response. In situ immunization is a strategy where immunomodulatory products such as pathogens are injected into one tumor site in order to trigger a systemic anti-tumor immune response. Of importance, pre-clinical rationale has demonstrated that combination of anti-CTLA4 therapy together with intra-tumoral (IT) oncolytic virus can overcome primary resistance to systemic anti-CTLA4 therapy. Pexastimogene Devacirepvec (Pexa-Vec) is one of the new vaccinia oncolytic viruses genetically modified to express GM-CSF. This new and innovative oncolytic virotherapy should therefore synergize with anti-CTLA4 therapy via virus-induced tumor cell death & tumor-antigen release, GM-CSF-induced recruitment/maturation/activation of antigen presenting cells, and anti-CTLA4-induced Treg blockade/depletion. Intra-tumoral delivery of immunostimulating agents should, therefore, provide lower toxicity of mAb targeting immune checkpoints. Of note, IT injections of GM-CSF-encoding oncolytic viruses have already been shown to induce immune-mediated tumor responses on local (injected) and distant (not injected) tumor sites. In solid injectable refractory/relapsing metastatic tumors, we make the hypothesis that the addition of Pexa-Vec to IT ipilimumab (anti-CTLA4 Ab) will overcome primary/secondary resistance to standard therapy and/or immunotherapy with a better in situ tumor antigen specific T-cell priming. Our proposal is to conduct a 2-part Phase I clinical trial in order to define the feasibility, the safety and the anti-tumor effects of intra-tumoral injections of ipilimumab in combination with the oncolytic virus Pexa-Vec. Dose escalation step will define the MTD and RP2D of that in situ immunization strategy. Expansion part will assess the anti-tumor effect of the combination.

DETAILED DESCRIPTION:
The study is a proof of concept, open label, multicentric, 2-parts, Phase I dose escalation trial. In dose selection part (any histological types except HCC), patients will be treated with an IT boost injection with Pexa-Vec (fixed dose of 1x109 pfu / injection ) alone at Week 1 followed by IT injections of Pexa-Vec + ipilimumab (up to 4 dose levels) at Weeks 3, 5 and 9. The dose escalation part will follow a classical 3+3 design. 3 to 6 patients will be enrolled at each DL (Dose Level) depending of the number of Dose Limiting Toxicity (DLT) observed. At the end of each DL cohort, a teleconference (Dose escalation meeting) will be organized with the sponsor, in order to select the dose for the next cohort. In Expansion cohorts ( up to 3 cohorts) patients will be treated with an IT boost injection with Pexa-Vec alone (fixed dose of 1x109 pfu / injection) at Week 1 followed by IT injections of Pexa-Vec + ipilimumab (RP2D) at Weeks 3, 5 and 9. In both parts, the treatment with both IMPs should be continued as per protocol until Withdrawal of consent, Disease progression as per irRC (immune related response criteria), General or specific changes in the patient's condition that render the patient unacceptable for further treatment in the judgment of the investigator, Pregnancy or Unacceptable adverse events(s) including DLTs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years at time of inform consent signature
* Histologically confirmed, advanced/metastatic solid tumor refractory or relapsing to/after standard therapy or the patient has refused or does not tolerate standard therapy. Any tumor types can be considered in Part A except hepatocellular carcinoma (HCC). In part B, tumor types may include melanoma, MSI-High colorectal carcinoma (CRC), head and neck tumors, gastric cancers, triple negative breast cancers and mesothelioma.
* Tumor status (as determined by radiology evaluation): At least one injectable site ≥2cm and ≤8 cm in diameter and one distant non-injected measurable site (target site).

NotaBene: for the DL5 and DL6, depending of the size of the injectable lesions, patients should present more than 1 injectable lesion (See Appendix 3). Of note, patients with only one injectable lesion with a diameter = 2 cm are not eligible for theses 2 DLs.

* PS ECOG 0 or 1
* Minimal wash-out period for prior anti-cancer regimens (i.e. chemotherapy, immunotherapy, or radiation therapy) > 3 weeks before Week 1 day 1.
* Resolution (i.e. ≤ Grade 1) of all toxicity related to prior anti-cancer treatment with exceptions of alopecia Grade 2, neuropathy Grade 2 and according to biological values presented in Criteria I8.
* No major surgery within 4 weeks prior Week 1 day 1
* Laboratory requirements:

  1. Absolute neutrophil count (ANC) ≥ 1 x 109/L
  2. Lymphocytes ≥1 x 109/L
  3. Platelets ≥ 100 x 109/L;
  4. Hemoglobin ≥ 90 g/L
  5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 3 x ULN (if patient exhibits liver metastasis, up to 5 x ULN acceptable) and total bilirubin ≤ 3mg/dL
  6. Serum creatinine ≤1.5 x ULN or creatinine clearance is ≥60 mL/min according to Cockcroft-Gault formula
  7. International normalized ratio (INR) ≤1.7
  8. Serum chemistries within normal limits (high or low) or Grade 1 (with exception of sodium, potassium, glucose, calcium, upon Investigator discretion)
* Life expectancy > 3 months
* Negative pregnancy test for women of child-bearing potential within 72 hours before Week 1 Day 1
* Men and women of reproductive potential must be willing to double barrier methods of contraception during the treatment period and for up to 6 weeks after last Pexa Vec administration.
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Known significant immunodeficiency due to underlying illness (e.g., HIV/AIDS) and/or immune-suppressive medication including systemic corticosteroids and/or blood CD4+ T-cells < 200/µL.
* History of auto-immunity or untreated wounds from infection or inflammatory skin conditions. Ancient auto-immunity with stable endocrine oral substitution and vitiligo could be considered eligible by investigators.
* Experience of a severe systemic reaction or side-effect as a result of a previous smallpox vaccination
* Ongoing severe inflammatory skin condition (as determined by the investigator) requiring medical treatment
* History of severe eczema (as determined by the investigator) requiring medical treatment
* Severe or unstable cardiac disease, including significant coronary artery disease requiring angioplasty or stenting within the preceding 12 months, unless well-controlled and on stable medical therapy for at least 3 months
* Medical conditions, per the investigator's judgment, that predispose the patient to untoward medical risk of tachycardia, or hypotension during or following treatment with Pexa-Vec
* Previous treatment with Pexa-Vec or other vaccinia vector based treatment
* Tumor tissue sample not available for biological studies (from the initial diagnosis and/or relapse) at time of inclusion
* History of allergic reactions attributed to one of the compound of ipilimumab or compound of similar composition (as per Yervoy SPC® - see Appendix 5)
* Hepatitis C virus therapy including interferon/pegylated interferon or ribavirin or by extension any other hepatitis C virus therapy that cannot be discontinued within 14 days prior to any Pexa Vec injection. Sponsor should be consulted if the patient is taking any other antiviral medications to determine eligibility and/or to determine wash-out duration.
* Significant bleeding event within the last 12 months that places the patient at risk for IT injection procedure based on Investigator assessment
* Anticoagulant or anti-platelet medication that cannot be interrupted prior to IT injections (as listed in the protocol).
* Inability to suspend treatment with anti-hypertensive medication (including but not limited to: diuretics, beta-blockers, angiotensin converting enzyme [ACE] inhibitors, aldosterone antagonists, etc.) for 48 hours prior to and 48 hours after each Pexa Vec injection.
* Prior malignancy except for the following: basal or squamous cell skin cancer, in situ cervical cancer, or other cancer adequately treated from which the patient has been disease-free for at least 3 years
* Active brain metastasis (treated and stable brain metastasis accepted).
* Any prior or planned organ transplant (e.g., liver transplant) or allogeneic hematopoietic stem cell transplantation.
* Pregnant or breastfeeding women
* Household contact exclusions for patients enrolled: Women who are pregnant or nursing an infant, Children < 1 year old, People with skin disease (e.g. eczema, atopic dermatitis and related diseases…), Immunocompromised hosts (severe deficiencies in cell-mediated immunity, including AIDS, organ transplant recipients, hematologic malignancies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Part A (dose selection part): Dose Limiting Toxicities (DLTs) | during the DLT assessment window (i.e. during the first 5 weeks of treatment)
  DLT is defined as the occurrence of any of the following events evaluated as related to study drugs and occurring during the first 5 weeks (Part A) of investigative treatment(s): any Grade ≥ 4 treatment related toxicity, any Grade≥ 3 treatment related toxicity lasting more than 7 days (except for flu-like symptoms that respond to standard therapies.), any Grade ≥ 3 treatment related acute immune related AE involving major end organs, Grade ≥ 3 injection site reaction, Any other study drug related toxicity considered significant enough to be qualified as DLT in the opinion of the investigators after discussion with the sponsor. Indeed, as a principle in this Phase I study, any toxicity that the investigator or the sponsor determines to be dose-limiting, regardless of the grade, may be considered as a DLT.
Part B (expansion cohort): The 3-month objective response rate (ORR) | 3 months of treatment
  The 3-month objective response rate is defined by the percentage of patients having complete response (CR) or partial response (PR) according to immune related Response Criteria (irRC).

SECONDARY OUTCOMES:
3-month objective response rate (ORR) | 3 months of treatment
  defined by the percentage of patients having complete response (CR) or partial response (PR) according to irRC (immune related Response Criteria) and to RECIST 1.1 criteria.
Best objective response rate | from the date of inclusion up to 12 months
  defined by the percentage of patients having complete response (CR) or partial response (PR) as best response at any time point according to irRC and to RECIST 1.1 criteria.
Disease Control Rate | from the date of inclusion up to 12 months
  defined by the rate of patients having complete response (CR), partial response (PR) or stable disease (SD) according to irRC and to RECIST 1.1 criteria.
Duration of response | from the time of first documented objective response (PR or CR according to irRC and to RECIST 1.1 criteria) until the first documented disease progression or death due to underlying cancer, assessed up to 12 months
ORR of injected and non injected lesions | from the date of inclusion up to 12 months
  OR defined as at least 50% decrease of tumor size
Progression Free Survival (PFS) | from the date of inclusion until the date of first documented event (progression, according to irRC and to RECIST 1.1 criteria, or death due to any cause),up to 12 months
  PFS will be estimated using Kaplan Meier method.
Time To progression (TTP) | from the date of inclusion until the date of first documented radiographic tumor progression, according to irRC and to RECIST 1.1 criteria, up to 12 months
  TTP does not include deaths
Overall Survival (OS) | from the time of inclusion, until the date of death due to any cause, up to 12 months
Adverse Events reporting | from the treatment start (Week1 Day 1), up to 12 months
  All AEs will be graded according to NCI-CTCAE, Version 4

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien MARABELLE, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (5):
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Léon Bérard, Lyon
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No